CLINICAL TRIAL: NCT06873529
Title: The Evaluation of Experiences of Women With Spinal Cord Injury Regarding Fertility, Contraception and Pregnancy
Brief Title: The Experiences of Women With Spinal Cord Injury Regarding Fertility, Contraception and Pregnancy
Status: Recruiting | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Örücü Atar, Associate professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: E-34215015
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injury
Keywords: fertility; contraception; pregnancy
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- spinal cord injury group: The evaluation of experiences of women with spinal cord injury regarding fertility, contraception and pregnancy

SUMMARY:
The aim of this study was to investigate the experiences of women with spinal cord injury regarding fertility, contraception and pregnancy.

DETAILED DESCRIPTION:
Although some studies exist in the literature on contraception and pregnancy in women with spinal cord injury, the data still remain insufficient.

The aim of this study was to investigate the experiences of women with spinal cord injury regarding fertility, contraception and pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-55
* Post-spinal cord injury period > 1 year

Exclusion Criteria:

* Having cognitive impairment

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with spinal cord injury who have been injured for at least 1 year
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation of experiences with fertility, contraception and pregnancy | through study completion, an average of one month
  The content of the survey used in the study was created by the research team after reviewing the current literature examining the parameters related to fertility, contraception and pregnancy in women with spinal cord injury. The survey consists closed-ended (e.g., use of a five-point Likert scale to assess whether spinal cord injury affects the decision to have children (Higher scores mean worse outcome)) and open-ended questions (e.g., What is the reason for choosing the contraceptive method used?)

CONTACTS AND LOCATIONS:
Overall Officials: Merve Örücü Atar, Principal Investigator — Ankara Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- Ankara Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)